CLINICAL TRIAL: NCT07357532
Title: Exploration of Treatment Strategies After Concurrent Chemoradiotherapy for Limited-stage Small Cell Lung Cancer (LS-SCLC) Guided by Molecular Residual Disease (MRD)
Brief Title: Exploration of Treatment Strategies After Concurrent Chemoradiotherapy for LS-SCLC Guided by MRD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ103
Record Dates: First submitted 2025-12-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: MRD-positive subjects will receive treatment with adebrelimab (anti-PD-L1) combined with apatinib (anti-angiogenic therapy),with close monitoring for disease progression.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD-positive group (Experimental): The specific dosing regimen is as follows:
  Adebrelimab: Intravenous infusion, 1200 mg, administered on Day 1 of each cycle, once every 3 weeks.
  Apatinib: Oral administration, 250 mg, once daily. Patients with limited-stage small cell lung cancer who have completed all radical chemoradiotherapy (prophylactic cranial irradiation is permitted) and test positive for MRD upon enrollment, without prior use of immune checkpoint inhibitors, will receive adebrelimab combined with apatinib according to the above dosing regimen. Treatment with adebrelimab and apatinib will continue, along with ongoing ctDNA monitoring. The above treatment regimen will be maintained until disease progression, intolerable toxicity, completion of two years of treatment, subject-initiated withdrawal, or investigator-determined discontinuation.
  Interventions: Drug: Adebrelimab Injection; Drug: Apatinib Mesylate Tablets

INTERVENTIONS:
Drug: Adebrelimab Injection — Patients with MRD Positive will receive adebrelimab (1200 mg, D1, Q3W) , followed by ctDNA monitoring every 2 months (Year 1) and every 3 months (Year 2).The above treatment regimen will be maintained until disease progression, intolerable toxicity, completion of two years of treatment, subject-initiated withdrawal, or investigator-determined discontinuation.
  Other Names: Ai Rui Li
Drug: Apatinib Mesylate Tablets — Apatinib Mesylate Tablets (250 mg, QD) , followed by ctDNA monitoring every 2 months (Year 1) and every 3 months (Year 2).The above treatment regimen will be maintained until disease progression, intolerable toxicity, completion of two years of treatment, subject-initiated withdrawal, or investigator-determined discontinuation.
  Other Names: Ai Tan

SUMMARY:
This study plans to enroll limited-stage small cell lung cancer (LS-SCLC) patients who have achieved disease control after concurrent chemoradiotherapy (cCRT). Tissue samples collected at initial diagnosis and serial peripheral blood samples obtained at multiple post-cCRT timepoints will be analyzed using targeted next-generation sequencing to investigate the correlation between molecular residual disease (MRD) status and tumor recurrence/metastasis. For patients with MRD-positive results, a therapeutic strategy combining immunotherapy with anti-angiogenic agents will be implemented with the aim of improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent; age >18 and <80 years;
2. Histologically or cytologically confirmed limited-stage small cell lung cancer (LS-SCLC);
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1;
4. Patients who have achieved disease stabilization after concurrent or sequential chemoradiotherapy;
5. Patients who had not received previous immune checkpoint inhibitor treatment;
6. Patients with MRD-positive status following concurrent chemoradiotherapy;
7. Willingness to provide clinical-pathological data, imaging studies, and other required materials for research purposes; compliance with follow-up procedures, including blood sample collection at predefined efficacy evaluation timepoints; and agreement to use the collected data for subsequent research analyses.

Exclusion Criteria:

1. Have other malignant tumors;
2. Autoimmune disorders that are not amenable to PD-L1 inhibitor therapy;
3. Prior exposure to other anti-angiogenic small molecule TKIs such as erlotinib or anti-angiogenic monoclonal antibodies such as bevacizumab (except locally infused bevacizumab); or participation in a clinical trial of another antineoplastic agent within 4 weeks prior to the first dose of ; or prior treatment with a paclitaxel;
4. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg despite optimal pharmacologic therapy);
5. Class II or greater myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc intervals ≥450 ms in men and ≥470 ms in women). According to NYHA criteria, grade III-IV cardiac insufficiency, or cardiac color ultrasound suggests that the left ventricular ejection fraction (LVEF) is <50% have had a myocardial infarction within 6 months prior to enrollment, New York Heart Association class II or higher heart failure, uncontrolled angina pectoris, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or ECG suggestive of acute ischemia or active conduction system abnormalities; (6) uncontrolled angina pectoris, uncontrolled severe ventricular arrhythmias, clinically significant pericardial disease, or ECG suggestive of acute ischemia or active conduction system abnormalities.
6. Uncontrolled co-morbidities including, but not limited to, poorly controlled diabetes mellitus, diabetic peripheral lesions , persistent infections, or psychiatric or social conditions that may interfere with the subject's ability to comply;
7. Abnormal coagulation (INR > 1.5 or Prothrombin Time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), hemorrhagic symptoms, or on thrombolytic or anticoagulant therapy;
8. Known hereditary or acquired bleeding and thrombotic disorders such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.;
9. Significant coughing up of fresh blood or hemoptysis of one-half teaspoon (2.5 ml) per day or more within 2 months prior to entry into the study ;
10. Failure to receive specified treatment or change in treatment regimen prior to disease progression;
11. Unable to cooperate with the study in accordance with the established clinical follow-up period;
12. Unable to accept or provide the specified means of efficacy assessment such as imaging.
13. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-09-26 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Negative conversion rate of MRD | MRD is assessed at 60-day intervals during the first year and 90-day intervals during the second year, until disease progression, study discontinuation for any reason, or completion of 2 years of follow-up, whichever occurs first.
  Patients with limited-stage small cell lung cancer (LS-SCLC) receive concurrent chemoradiotherapy in accordance with standard diagnostic and treatment guidelines. Patients who are MRD-positive after completion of concurrent chemoradiotherapy and have not previously been treated with immune checkpoint inhibitors are screened and enrolled to receive the investigational treatment regimen. We then calculate the proportion of patients whose MRD status converts from positive to negative following treatment.

SECONDARY OUTCOMES:
PFS | Imaging assessments are performed every 3 months. After each assessment, treatment response is evaluated by senior experts according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. The maximum follow-up duration is 2 years.
  Progression-Free Survival (PFS) is defined as the time interval from randomization (or treatment initiation in single-arm studies) to the first occurrence of either: Radiographically or pathologically confirmed disease progression（RECIST1.1）, or Death from any cause; whichever is observed first.
OS | Imaging assessments are performed every 3 months. After each assessment, treatment response is evaluated by senior experts according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. The maximum follow-up duration is 2 years.
  Overall Survival (OS) is defined as the time interval from randomization (or treatment initiation in single-arm studies) to death from any cause.
Time to conversion to MRD negativity | MRD is assessed at 60-day intervals during the first year and 90-day intervals during the second year, until disease progression, study discontinuation for any reason, or completion of 2 years of follow-up, whichever occurs first.
  Patients with limited-stage small cell lung cancer (LS-SCLC) receive concurrent chemoradiotherapy in accordance with standard diagnostic and treatment guidelines. Patients who are MRD-positive after concurrent chemoradiotherapy and have no prior exposure to immune checkpoint inhibitors are screened and enrolled to receive the investigational treatment regimen. The time required for MRD conversion from positive to negative following treatment is calculated, measured in days.
Duration of negative conversion after medication in MRD-positive patients | MRD is assessed at 60-day intervals during the first year and 90-day intervals during the second year, until disease progression, study discontinuation for any reason, or completion of 2 years of follow-up, whichever occurs first.
  Patients with limited-stage small cell lung cancer (LS-SCLC) receive concurrent chemoradiotherapy in accordance with standard diagnostic and treatment guidelines. Patients who are MRD-positive after concurrent chemoradiotherapy and have no prior exposure to immune checkpoint inhibitors are screened and enrolled to receive the investigational treatment regimen. The duration of MRD negativity after treatment-defined as the time from conversion to MRD-negative status to subsequent reversion to MRD-positive status, if applicable-is calculated and measured in days.

OTHER OUTCOMES:
Dynamic Changes in Absolute Counts and Activation Status of Peripheral Blood Lymphocyte Subsets | It is assessed at 60-day intervals during the first year and 90-day intervals during the second year, until disease progression, study discontinuation for any reason, or completion of 2 years of follow-up, whichever occurs first.
  Patients with limited-stage small cell lung cancer (LS-SCLC) receive concurrent chemoradiotherapy in accordance with standard diagnostic and treatment guidelines. Patients who are MRD-positive after concurrent chemoradiotherapy and have no prior exposure to immune checkpoint inhibitors are screened and enrolled to receive the investigational treatment regimen. Changes in the counts and functional activity of peripheral blood lymphocyte subsets are then evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhao, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No